CLINICAL TRIAL: NCT05822843
Title: A Phase I, Open Label, Multiple Dose, Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics and Antitumor Activities of Anti-BAFFR mAb(Monoclonal Antibody), ESG206 in Subjects With B-cell Lymphoid Malignancies
Brief Title: A Phase 1 Study of ESG206 in Adult Subjects With B-cell Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Escugen Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ESG206-102
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: B-cell Lymphoid Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ESG206 dose level 1 (Experimental): ESG206 will be administered intravenously at dose level 1 every two weeks in a 28-day cycle
  Interventions: Drug: ESG206
- ESG206 dose level 2 (Experimental): ESG206 will be administered intravenously at dose level 1 every two weeks in a 28-day cycle
  Interventions: Drug: ESG206
- ESG206 dose level 3 (Experimental): ESG206 will be administered intravenously at dose level 1 every two weeks in a 28-day cycle
  Interventions: Drug: ESG206
- ESG206 dose level 4 (Experimental): ESG206 will be administered intravenously at dose level 1 every two weeks in a 28-day cycle
  Interventions: Drug: ESG206

INTERVENTIONS:
Drug: ESG206 — Administered via intravenous (IV) infusion

SUMMARY:
This is a phase I, multicenter, open label, sequential-cohort, dose escalation study of ESG206. The purpose is to evaluate the clinical safety, tolerability, PK (pharmacokinetics), and preliminary efficacy and to establish the MTD (maximum tolerated dose), if any, and RP2D (recommended phaseII dose) of ESG206 in adult subjects with B lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for the trial.
* Male or female and at least 18 years of age.
* Subjects must have a histologically confirmed (or documented), incurable B-cell hematologic malignancy that had progressed despite standard of care therapy and for which there was no alternative therapy of proven benefit or no effective standard therapy is available or tolerable.
* Measurable or evaluable Disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subject must have adequate organ function.

Exclusion Criteria:

* Has had prior chemotherapy, targeted therapy, immunotherapy or any other agents used as systemic treatment for cancer, within 14 days before first dosing.
* Had major surgery within 4 weeks before first dosing.
* Had undergone an autologous stem cell transplant within 100 days before first dosing.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, or renal disease).
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the investigational product or excipients.
* Pregnant or breastfeeding women.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Any Treatment Emergent Adverse Events | First dose date up to last dose plus 30 days
  Treatment-emergent adverse events (TEAEs) were defined as: Any adverse event (AE) that happens after treatment initiation, or AE that was present at time of treatment initiation but worsened after treatment initiation, or AE that was present and resolved prior to treatment and reappeared after treatment initiation after the start of study drug through 30 days after the last dose of study drug. The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events.

SECONDARY OUTCOMES:
Cmax | Up to 20 months
  Maximum observed plasma concentration
AUC0-inf | Up to 20 months
  Area under the serum concentration time curve (AUC) from time 0 extrapolated to infinity
Tmax | Up to 20 months
  Time to maximum plasma concentration
T1/2 | Up to 20 months
  Half-life
Overall Response Rate (ORR) | Up to 20 months
  Defined as complete response (CR) + partial response (PR)
Progression-free Survival (PFS) | Up to 20 months
  Defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression or death from any cause
ADA | Up to 20 months
  Incidence of anti-drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No